CLINICAL TRIAL: NCT01597804
Title: A "Bathing Bundle" Regimen to Reduce the Risk of Gynecological Surgical Site Infection
Brief Title: Bathing Bundle Regimen in Reducing Gynecological Surgical Site Infection in Patients Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: I 189910; NCI-2012-00273 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 189910 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Malignant Female Reproductive System Neoplasm
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Supportive care ("Bathing Bundle") (Experimental): Patients undergo preoperative preparation with the "Bathing Bundle" comprising CHG 4% skin prep solution and disposable wash cloths to bathe or shower with the night before and morning of surgery.
  Interventions: Procedure: Infection Prophylaxis and Management

INTERVENTIONS:
Procedure: Infection Prophylaxis and Management — Undergo preoperative preparation with the "Bathing Bundle"
  Other Names: Infectious Diseases / Treatment, General; infectious diseases treatment; management, infection prophylaxis; Treatment of Infectious Disease

SUMMARY:
This pilot clinical trial studies bathing bundle regimen in reducing gynecological surgical site infection in patients undergoing surgery. A bathing bundle regimen may reduce the risk of wound infection, extended length of hospital stay, readmission into the hospital, and the overall healthcare costs in patients undergoing surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate whether gynecology surgical patients using a Bathing Bundle using chlorhexidine gluconate (CHG) 4% skin prep solution (Intervention Group A) have a lower incidence of surgical site infection (SSI) than patients treated with the current standard of care (patient's choice of antibacterial soap). Standard of care results will be based on historical information gathered on Roswell Park Cancer Institute (RPCI) gynecology (GYN) patients prior to July 1, 2010 (Historical Control Group B).

OUTLINE:

Patients undergo preoperative preparation with the "Bathing Bundle" comprising CHG 4% skin prep solution and disposable wash cloths to bathe or shower with the night before and morning of surgery.

After completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* GYN surgical patients scheduled for abdominal surgery

Exclusion Criteria:

* Patients with known hypersensitivity to chlorhexidine
* GYN non-surgical patients or surgical patients that will not have an abdominal incision (i.e. vaginal procedures)

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2011-04; Primary Completion 2014-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Presence of a site infection, compared with historical SSI rates among RPCI GYN surgery patients treated with the standard of care before July 1, 2010 | Within 30 days following surgery
  Assessed using Fisher's exact test. This primary analysis will be supplemented by logistic regression modeling for the probability of an SSI given the bathing regimen used, controlling for compliance and other patient characteristics of interest. The pre- and post intervention patient samples will be compared on various demographic, health behavior, and disease characteristics. Descriptive statistics and various graphical displays will be provided as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Barbra Dodds, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States